CLINICAL TRIAL: NCT04816409
Title: Effect of Neuro Developmental Therapy to Improve Postural Reactions and Motor Milestones in Infants With Down Syndrome
Brief Title: Effect of Neuro Developmental Therapy in Infants With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/Lhr/19/1010 Raneem sajjad
Record Dates: First submitted 2021-03-24; First posted 2021-03-25 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Children; Gross motor function; Neurodevelopmental treatment; Rehabilitation; Milestones; Postural reactions
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (Neurodevelopmental therapy) (Experimental): Starting Posture Start and evaluate the supreme effective posture to move from(usually straight) Reassemble to mid plane (head/trunk)
  •Neutral position of body Identify the Missing Components Detect starting posture and compare to normal.
  Neurodevelopmental therapy application :
  Tonic postural extensor muscle strengthening:
  Push-pull scooter board games contrary to resistive tubing strips.
  Developmental movement patterns training:
  Obstacle crawl, hold swing's ropes in kneeling anhalf kneeling position, throw balls to aim kneeling and standing position. Manual Cues .Use hands on key points of control to assist normal posture, movement and prevent abnormal posture and movement. Balance and corrective reactions was established by means of ball and tilt board after the development of the skill of sustaining exercise positions in children.4. Ambulation training, suitable to the motor
  Interventions: Other: Neurodevelopmental therapy
- Conventional treatment (Active Comparator): Range of motion and Resistance training Linear actions are used to regularize extensor muscle tone (Neck extensors, back extensors hip extensors, knee extensors).(49) Postural control exercises Bouncing on gym ball in sitting, kneeling, or standing Linear swinging using a platform and swing, glider, hammock, and barrel; swinging in the kneeling, standing, sitting,
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: conventional therapy — Range of motion and Resistance training Linear actions are used to regularize extensor muscle tone (Neck extensors, back extensors hip extensors, knee extensors).(49) Postural control exercises Bouncing on gym ball in sitting, kneeling, or standing
  - Linear swinging using a platform and swing, glider, hammock, and barrel; swinging in the kneeling, standing, sitting,
  Arms: Conventional treatment
Other: Neurodevelopmental therapy — Starting Posture
  * Start and evaluate the supreme effective posture to move from(usually straight)
  * Reassemble to mid plane (head/trunk)
  * Neutral position of body (47) Identify the Missing Components Detect starting posture and compare to normal.(47)
  Neurodevelopmental therapy application :
  Tonic postural extensor muscle strengthening:
  Push-pull scooter board games contrary to resistive tubing strips.(48) 2. Developmental movement patterns training: Obstacle crawl, hold swing's ropes in kneeling and half kneeling position, throw balls to aim kneeling and standing position. Manual Cues .Use hands on key points of control to assist normal posture, movement and prevent abnormal posture and movement. Balance and corrective reactions was established by means of ball and tilt board after the development of the skill of
  li
  Arms: (Neurodevelopmental therapy)

SUMMARY:
Neurodevelopmental treatments are a progressive therapeutic method experienced thru qualified therapists for the improvement in affected ones. The most important trial in Down syndrome children is motor milestones and postural reactions to develop on time.

Neurodevelopmental therapy is applied to accurate atypical postural tone and to enable further regular motion for execution of presentation of abilities. Objective: To determine the effects of Neuro Developmental therapy in improving postural reaction and motor milestones in infants with Down syndrome.

DETAILED DESCRIPTION:
This study was a randomized trial design. This study was conducted in Rehab Care Physiotherapy Department. 20 Children with Down syndrome meeting the predetermined inclusive and exclusive criteria were arbitrarily allocated into dual batches through convenient sampling technique. The first batch which was the experimental group was given Neurodevelopmental therapy and the duration of the treatment comprised of 1.5 hour, three days a week for 6 weeks. The second group which was the control group received conventional therapy and the period of the ministrations comprised of 1 hour, with 10 repetition 3 sets for each muscle three days a week for 1.5 months, Pre-assessment and post-assessment was evaluated through Gross motor function-88. Recorded values were analyzed through SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Trisomy 21 by genetic karyotype.
* Down syndrome children with delayed milestone.
* Definite identification of Down syndrome by neurologist.
* Children having the average birth weight above 2.500 grams and average birth length above 49.52 cm.
* Laxity, low muscle tone and psychomotor development deficits

Exclusion Criteria:

* Infants with Heart Defect.
* Seizure.
* Critical orthopedic difficulties or deformities (hip instability, patellar instability, foot deformity).
* Unrestrained thyroid conflicts.
* Perilabour asphyxia (Apgar of minutes 1 and 5 equal to or less than 7).
* Critical optical or acoustic disorders.
* Mass below the 3rd percentage of Down syndrome

Ages: 5 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
Gross Motor Function Measure-88(GMFM-88) | 2 months
  The GMFM-88 is the original 88-item measure. Items span the spectrum of gross motor activities in five dimensions. ... The GMFM-66 is a 66 item subset of the original 88 items identified through Rasch analysis to best describe the gross motor function of children with cerebral palsy of varying abilities.

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Binash afzal, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angsupaisal M, Dijkstra LJ, la Bastide-van Gemert S, van Hoorn JF, Burger K, Maathuis CGB, Hadders-Algra M. Best seating condition in children with spastic cerebral palsy: One type does not fit all. Res Dev Disabil. 2017 Dec;71:42-52. doi: 10.1016/j.ridd.2017.09.016. Epub 2017 Oct 5. PMID 28987971
- [Background] Valentin-Gudiol M, Mattern-Baxter K, Girabent-Farres M, Bagur-Calafat C, Hadders-Algra M, Angulo-Barroso RM. Treadmill interventions in children under six years of age at risk of neuromotor delay. Cochrane Database Syst Rev. 2017 Jul 29;7(7):CD009242. doi: 10.1002/14651858.CD009242.pub3. PMID 28755534
- [Background] Mura G, Carta MG, Sancassiani F, Machado S, Prosperini L. Active exergames to improve cognitive functioning in neurological disabilities: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Jun;54(3):450-462. doi: 10.23736/S1973-9087.17.04680-9. Epub 2017 Oct 25. PMID 29072042
- [Background] O'Callaghan FJ, Edwards SW, Alber FD, Hancock E, Johnson AL, Kennedy CR, Likeman M, Lux AL, Mackay M, Mallick AA, Newton RW, Nolan M, Pressler R, Rating D, Schmitt B, Verity CM, Osborne JP; participating investigators. Safety and effectiveness of hormonal treatment versus hormonal treatment with vigabatrin for infantile spasms (ICISS): a randomised, multicentre, open-label trial. Lancet Neurol. 2017 Jan;16(1):33-42. doi: 10.1016/S1474-4422(16)30294-0. Epub 2016 Nov 10. PMID 27838190
- [Background] Armstrong D, Said RR. Outcomes of High-Dose Steroid Therapy for Infantile Spasms in Children With Trisomy 21. J Child Neurol. 2019 Oct;34(11):646-652. doi: 10.1177/0883073819850650. Epub 2019 May 22. PMID 31113280
- [Background] Alsakhawi RS, Elshafey MA. Effect of Core Stability Exercises and Treadmill Training on Balance in Children with Down Syndrome: Randomized Controlled Trial. Adv Ther. 2019 Sep;36(9):2364-2373. doi: 10.1007/s12325-019-01024-2. Epub 2019 Jul 12. PMID 31301057
- [Background] Savardi A, Borgogno M, Narducci R, La Sala G, Ortega JA, Summa M, Armirotti A, Bertorelli R, Contestabile A, De Vivo M, Cancedda L. Discovery of a Small Molecule Drug Candidate for Selective NKCC1 Inhibition in Brain Disorders. Chem. 2020 Aug 6;6(8):2073-2096. doi: 10.1016/j.chempr.2020.06.017. PMID 32818158